CLINICAL TRIAL: NCT05186025
Title: A Long-term, Prospective, Open, Multi-centre, Non-interventional Study to Evaluate the Effectiveness After Treatment With TA Bäume Top (Trees) and TA Gräser Top (Grass) Following a Perennial Posology in Children and Adults, as Well as Proofing the Non-inferiority of Children Compared to Adults
Brief Title: Tyrosine Allergoid Paediatric and Adult Study
Status: Active, not recruiting | Type: Observational
Sponsor: Allergy Therapeutics (Industry)
Collaborators: Bencard Allergie GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: TAPAS
Record Dates: First submitted 2021-10-20; First posted 2022-01-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Allergic Rhinitis Due to Pollen; Allergic Conjunctivitis; Allergic Asthma
Keywords: Allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adults: adult patients aged ≥ 18 with rhinitis, conjunctivitis and/or mild to moderate bronchial asthma, caused by an IgE-mediated allergy to grass/rye or tree pollen; who are treated with MATA grass or MATA trees as part of their routine medical care
  Interventions: Drug: MATA trees or MATA grass
- Children: children aged from >5 to 17 years with rhinitis, conjunctivitis and/or mild to moderate bronchial asthma, caused by an IgE-mediated allergy to grass/rye or tree pollen; who are treated with MATA grass or MATA trees as part of their routine medical care
  Interventions: Drug: MATA trees or MATA grass

INTERVENTIONS:
Drug: MATA trees or MATA grass — Glutaraldehyde-modified and MCT® (MicroCrystalline Tyrosine)-adsorbed allergoids
  Other Names: TA Gräser; TA Bäume

SUMMARY:
The primary objective of this 5-year study is to demonstrate non-inferiority of children compared to adults by exploring long-term effectiveness after treatment with TA Bäume (trees) and TA Gräser (grass) following a perennial posology.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 5 years of age who are treated with TA Gräser top or TA Bäume top due to rhinitis, conjunctivitis and/or mild to moderate bronchial asthma, which are caused by an IgE-mediated allergy to grass and rye pollen or birch, alder and hazel pollen according to the respective SmPC.
* Patients will only be included in this study after the decision on the treatment has been made.

Exclusion Criteria:

* History of allergen-specific immunotherapy (SIT) for trees or grass within the last 5 years
* If it´s intended to treat the patient with only a preseasonal therapy
* A patient should also not be included in the presence of any of the conditions listed in the respective SmPC

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults, adolescents and children from the age of 5 on, who are going to be treated with TA Bäume or TA Gräser.
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
change in the combined symptom medication score (CSMS) | once a year for 5 years
  The primary endpoint is the change in the total combined symptom medication score (CSMS) during the entire study period, determined from the rhinoconjunctivitis daily symptom score (dSS) and rhinoconjunctivitis daily medication score (dMS), averaged over the respective peak pollen season

SECONDARY OUTCOMES:
rhinoconjunctivitis daily medication score | once a year for 5 years
  the changes in use of daily anti-allergic medication needed, averaged over the respective peak pollen season
rhinoconjunctivitis daily symptom score | once a year for 5 years
  allergic symptoms and severity will be self-recorded by the subject in an eDiary on a daily basis during the pollen season, averaged over the respective peak pollen season
Rhinoconjunctivitis Quality of Life | twice a year for 5 years
  The change in quality of life as assessed by the standardised Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ(s))
Rhinitis Control | twice a year for 5 years
  change in symptom control of rhinitis assessed by Rhinitis Control Assessment Test (RCAT)
Asthma Control | twice a year for 5 years
  The change of asthma control in asthmatic patients assessed by the (Childhood) Asthma Control Test (C-ACT/ACT)
Incidence of Treatment-Emergent Adverse Events (safety and tolerability) | all year for 3 years
  frequency and severity of Treatment-Emergent adverse events
treatment satisfaction | once after 3 years and once after 5 years
  directly assessed by the physician (questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Moesges, Prof., Principal Investigator — ClinCompetence Cologne GmbH
Locations (1):
- Universitätsklinikum Augsburg, Augsburg, Germany